CLINICAL TRIAL: NCT07350551
Title: Pediatric Epilepsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Angela Price, Clinical Associate Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU20251324
Record Dates: First submitted 2025-12-16; First posted 2026-01-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Epilepsy Intractable
Keywords: Epilepsy; Decision-making; Cognitive control; Memory; Depth Electrode; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; ADHD (Attention-Deficit/Hyperactivity Disorder); Cognitive development
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Arm (Cognitive testing) (Experimental): All participants will undergo series of cognitive task testing with some involving tasks contexts such as incentives, cognitive loads, presence of a neutral image or verbal instructions being changed at different times and components where subjects learn and memorize facts and make decisions using such knowledge to obtain Behavioral and Neuronal Recordings of change in task performance.
  Interventions: Behavioral: Cedrus RB series response pad; Adtech Behnke-Fried micro-electrodes; Neuralynx or Blackrock electrophysiology system; Blackrock Cerestim or Natus Nicolet stimulator

INTERVENTIONS:
Behavioral: Cedrus RB series response pad; Adtech Behnke-Fried micro-electrodes; Neuralynx or Blackrock electrophysiology system; Blackrock Cerestim or Natus Nicolet stimulator — Devices listed are components of a single intervention that includes: Record patient responses (Cedrus RB series response boxes), record neuronal activity (Neuralynx or BlackRock) from electrodes (Adtech Behnke-Fried), apply intermittent electrical stimulation (Blackrock Cerestim, Natus Nicolet; parameters consistent with safe ranges across reported studies)

SUMMARY:
The purpose of the research is to better understand how the human brain accomplishes the basic cognitive tasks of learning new information, recalling stored information, making decisions or choices about presented information and self-control. These investigations are critical to better understand human cognition and to design treatments for disorders of learning, memory, decision making and cognitive control.

DETAILED DESCRIPTION:
The knowledge gained from these experiments furthers the understanding of the brain's electrical activity and its relation to epilepsy and to human cognition. This increased knowledge base may lead to insights regarding better treatments for cognitive deficits and to improve epilepsy surgery and other therapies for seizure disorders. Functional mapping is an important element of planning for resection surgery because it enables the surgeon to avoid the resection of brain regions that could be especially crucial to cognitive function. By uncovering the iEEG (Intracranial Electroencephalography) signatures of memory function, functional mapping may be improved, and the risk of post-surgical cognitive impairment following resection could be reduced.

Hypotheses being tested (conceptual: see "Data Analysis" section for specific hypotheses) The study team hypothesizes that specific electrophysiological correlates of successful memory encoding can be identified from the local field potentials recorded from subdural and intracranial depth electrodes. The study team believes that an analysis of local field potentials can provide insight into the organization of functional brain networks involved in memory encoding and retrieval.

Theta Oscillations and Behavior in Rodents Scientists have theorized, based predominantly on research in rodents, that brain oscillations - cyclic changes in the electrical activity recorded from electrodes - play a fundamental role in memory function. In particular, theories of the role of oscillations in cognitive function have focused on a slow rhythm in the 3- to 12-Hz frequency range, which is termed the theta rhythm. These slow oscillations appear prominently in recordings from the rat hippocampus, a region known to be important in learning and memory function across species.

The theta rhythm increases during movement, orienting, a simple form of learning called conditioning, short-term memory, and spatial learning. In addition, the phase within the theta cycle (i.e., whether you are at the peak or the trough of the wave) is important for memory function. When information is presented to the animal at the peak of the theta cycle, learning is enhanced. Although most research in the rat has focused on the hippocampal theta rhythm, theta oscillations have also been found in numerous other brain regions in both rats and other animals, suggesting that they play a very general role in the way brain networks operate.

Human Intracranial Recordings Although one can crudely measure the human brain's electrical signals by recording from the scalp, the ability to actually observe and measure oscillations generated in local regions of the brain requires recordings taken from electrodes implanted in the brain (i.e., invasive EEG, or iEEG recording). Such iEEG recordings are often clinically required in the surgical treatment of severe medication-resistant epilepsy (i.e., seizure disorders that are not controlled by standard drug therapies). The location of electrodes is selected for each patient on the basis of clinical needs. This often includes electrodes in the mesial temporal lobe, including the hippocampus and entorhinal cortex along with cortical surface electrodes. At UTSW (UT Southwestern Medical Center), the use of stereo encephalography provides the unique opportunity to record from multiple deep brain locations and examine properties of electrical activity suggesting communication between these areas.

iEEG recordings taken during treatment for intractable epilepsy (as described above) have already been used to greatly enhance our knowledge of the physiology of human cognition. First, iEEG recordings sample from much smaller brain volumes than scalp-recorded EEG or magnetoencephalographic (MEG) signals, are not subject to distortions produced by the human skull, and are relatively impervious to movement artifacts because of their high signal-to-noise ratio. iEEG recordings also offer far better temporal resolution than functional magnetic resonance imaging (fMRI).

ELIGIBILITY:
Inclusion Criteria:

* Candidates will be those who are admitted to the Epilepsy Monitoring Unit and are able to participate in a pre-operative evaluation using depth intracranial electrodes. The candidacy is determined independently by the patient's treating physician as part of the patient's routine medical care.
* Patients have drug-intractable epilepsy undergoing invasive monitoring in the EMU.

Exclusion Criteria:

* Determination by clinicians and investigators that a patient is unable to complete the behavioral tasks required for the protocol due to either cognitive limits, psychological limits, or pain.

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2031-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Intracranial electroencephalography (iEEG) power in the theta band | 5 years
  Time-frequency analyses of iEEG data during decision making
iEEG high-gamma activity | 5 years
  Time-frequency analyses of iEEG data during decision making
iEEG theta-gamma phase-amplitude coupling | 5 years
  Time-frequency analyses of iEEG data during decision making
Decision-making (firing rates) | 5 years
  Firing rates of neurons (measured in spikes per second) in the frontal and temporal lobes during a decision-making process.
Behavioral accuracy (neuromodulation) | 5 years
  Measure task accuracy observed in response to small pulses delivered by electrical stimulation during cognitive testing.
Reaction times (neuromodulation) | 5 years
  Measure reaction times on task observed in response to small pulses delivered by electrical stimulation during cognitive testing.
Firing rate (neuromodulation) | 5 years
  Measure firing rates of neurons (measured in amplitude across frequency of the bandwidths) in response to pulses of electrical activity during cognitive testing.

CONTACTS AND LOCATIONS:
Overall Officials: Angela V Price, M.D., Principal Investigator — UT Southwestern
Locations (1):
- Children's Medical Center Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No